CLINICAL TRIAL: NCT00768755
Title: Randomized Phase 2 Study Of Cisplatin/Pemetrexed With Or Without Axitinib (AG-013736) As First-Line Treatment For Patients With Non-Squamous Non-Small Cell Lung Cancer
Brief Title: Evaluation Of The Efficacy Of The Combination Of Axitinib With Pemetrexed And Cisplatin In The Treatment Of Non-Squamous Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4061039
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Results first posted 2012-03-30 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Carcinoma, Non-Small Cell Lung
Keywords: non-squamous NSCLC; axitinib; pemetrexed/cisplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Axitinib; Drug Therapy; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- I (Experimental): Axitinib (continuous) + Pemetrexed(500mg/m2)/Cisplatin(75mg/m2) x max 6 cycles followed by axitinib maintenance
  Interventions: Drug: axitinib
- II (Experimental): Axitinib (modified) + Pemetrexed(500mg/m2)/Cisplatin(75mg/m2) x max 6 cycles followed by axitinib maintenance
  Interventions: Drug: axitinib
- III (Active Comparator): pemetrexed and cisplatin
  Interventions: Drug: chemotherapy
- IV (Experimental): Axitinib interrupted before each chemo cycle (Pemetrexed(500mg/m2)/Cisplatin(75mg/m2) x max 6 cycles followed by axitinib maintenance
  Interventions: Drug: axitinib
- V (Active Comparator): pemetrexed and cisplatin
  Interventions: Drug: chemotherapy

INTERVENTIONS:
Drug: axitinib — 5mg BID po up to max 10mg BID po
  Other Names: AG-013736
  Arms: I
Drug: axitinib — 5mg BID po up to max 10mg BID po paused for 3 days before each cycle of concomitant chemotherapy
  Other Names: AG-013736
  Arms: II
Drug: chemotherapy — Pemetrexed(500mg/m2)/Cisplatin(75mg/m2) x max 6 cycles
  Other Names: alimta
  Arms: III
Drug: axitinib — 5mg BID po up to max 10mg BID po paused before each concomitant chemotherapy
  Arms: IV
Drug: chemotherapy — Pemetrexed(500mg/m2)/Cisplatin(75mg/m2) x max 6 cycles
  Other Names: alimta
  Arms: V

SUMMARY:
AG-013736 (axitinib) in combination with cisplatin and pemetrexed will be evaluated as first-line treatment of patients with locally advanced, recurrent, or metastatic non-squamous, non small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of adeno-, large cell or bronchioalveolar non-small cell lung cancer
* Cytologic specimens for diagnosis or for cell type classification must have been obtained from bronchial brushings or washings or from needle aspiration of a defined lesion. Sputum cytology alone will not be acceptable for diagnosis or for cell type classification.
* Patients with mixed NSCLC with predominantly squamous cell carcinoma should be classified as squamous and thus do not qualify for this study.
* Stage IIIB with malignant effusion (with cytologic confirmation of malignant pleural or pericardial effusion), Stage IV, or recurrent disease after definitive loco-regional therapy.
* Candidate for primary treatment with cisplatin and pemetrexed

Exclusion Criteria:

* Any histological/cytological evidence of predominantly squamous NSCLC.
* Small cell or carcinoid lung cancer patients are also ineligible.
* NSCLC that cannot be classified as one of the eligible histologies (adenocarcinoma, large cell or bronchioalveolar).
* Prior systemic therapy for Stage IIIB (with malignant effusion), Stage IV, or recurrent NSCLC. (Prior treatment with systemic therapy as adjuvant chemotherapy or in conjunction with radiotherapy for Stage II or III NSCLC is permitted if the last dose of chemotherapy was completed 12 months or more prior to randomization).
* Prior treatment with a VEGF or VEGFR inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2009-01; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (45):
- United States (11):
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Macon, Georgia
  - Pfizer Investigational Site, Marietta, Georgia
  - Pfizer Investigational Site, Sandy Springs, Georgia
  - Pfizer Investigational Site, Bloomington, Illinois
  - Pfizer Investigational Site, Peoria, Illinois
  - Pfizer Investigational Site, Hershey, Pennsylvania
  - Pfizer Investigational Site, West Reading, Pennsylvania
  - Pfizer Investigational Site, East Providence, Rhode Island
- Italy (3):
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Lido Di Camaiore (LU)
  - Pfizer Investigational Site, Orbassano (TO)
- Pfizer Investigational Site, Sunto-gun, Shizuoka, Japan
- Poland (6):
  - Pfizer Investigational Site, Lubin
  - Pfizer Investigational Site, Otwock
  - Pfizer Investigational Site, Piła
  - Pfizer Investigational Site, Poznan
  - Pfizer Investigational Site, Prabuty
  - Pfizer Investigational Site, Warsaw
- Romania (2):
  - Pfizer Investigational Site, Bacau, Bacău
  - Pfizer Investigational Site, Iași, Iaşi
- Russia (3):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Pyatigorsk
  - Pfizer Investigational Site, Saint Petersburg
- Spain (5):
  - Pfizer Investigational Site, Terrassa, Barcelona
  - Pfizer Investigational Site, Castellon, Castellon
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Palma de Mallorca, Palma de Mallorca
  - Pfizer Investigational Site, Seville, Sevilla
- Switzerland (3):
  - Pfizer Investigational Site, Basel
  - Pfizer Investigational Site, Bruderholz
  - Pfizer Investigational Site, Liestal
- Taiwan (2):
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Taipei
- Ukraine (2):
  - Pfizer Investigational Site, Dnipropetrovsk
  - Pfizer Investigational Site, Kyiv
- United Kingdom (7):
  - Pfizer Investigational Site, Romford, Essex
  - Pfizer Investigational Site, Northwood, Middlesex
  - Pfizer Investigational Site, Bournemouth
  - Pfizer Investigational Site, Brighton
  - Pfizer Investigational Site, Dundee
  - Pfizer Investigational Site, Middlesex
  - Pfizer Investigational Site, Poole

REFERENCES:
- [Derived] Belani CP, Yamamoto N, Bondarenko IM, Poltoratskiy A, Novello S, Tang J, Bycott P, Niethammer AG, Ingrosso A, Kim S, Scagliotti GV. Randomized phase II study of pemetrexed/cisplatin with or without axitinib for non-squamous non-small-cell lung cancer. BMC Cancer. 2014 Apr 25;14:290. doi: 10.1186/1471-2407-14-290. PMID 24766732
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061039

RESULTS

PARTICIPANT FLOW:
Groups:
- Axitinib + Pemetrexed/Cisplatin (Phase 1): Lead-in axitinib (AG-013736) tablet at a starting dose of 5 milligram (mg) orally twice daily (BID) from Day -5, -4 or -3 till Day 18 of Cycle 1 then continuously from Day 3 of Cycle 2 along with pemetrexed 500 milligram per square meter (mg/m^2) infusion and cisplatin 75 mg/m^2 infusion over a 2 hour period on Day 1 of each cycle up to 6 cycles of length 21 days each in chemotherapy phase and axitinib (AG-013736) tablet 5 mg orally BID in single-agent maintenance phase. Treatment was continued until progression of disease, unmanageable adverse events (AEs), or participant withdrawal.
- Axitinib (Continuous) + Pemetrexed/Cisplatin (Phase 2): Axitinib (AG-013736) tablet at a starting dose of 5 mg orally BID along with pemetrexed 500 mg/m^2 infusion and cisplatin 75 mg/m^2 infusion over a 2 hour period on Day 1 of each cycle up to 6 cycles of length 21 days each in chemotherapy phase and axitinib (AG-013736) tablet 5 mg orally BID in single-agent maintenance phase. Treatment was continued until progression of disease, unmanageable AEs, or participant withdrawal.
- Axitinib (Modified) + Pemetrexed/Cisplatin (Phase 2): Axitinib (AG-013736) tablet at a starting dose of 5 mg orally BID from Day 2-19 in cycles of chemotherapy phase, except the last cycle, where axitinib (AG-013736) was administered on Day 2-21 along with pemetrexed 500 mg/m^2 infusion and cisplatin 75 mg/m^2 infusion over a 2 hour period on Day 1 of each cycle up to 6 cycles of length 21 days each in chemotherapy phase and axitinib (AG-013736) tablet 5 mg orally BID in single-agent maintenance phase. Treatment was continued until progression of disease, unmanageable AEs, or participant withdrawal.
- Pemetrexed/Cisplatin (Phase 2): Pemetrexed 500 mg/m^2 infusion and cisplatin 75 mg/m^2 infusion over a 2 hour period on Day 1 of each cycle up to 6 cycles of length 21 days each in chemotherapy phase. Treatment was continued until progression of disease, unmanageable AEs, or participant withdrawal.
Period: Phase 1
Arm/Group | Axitinib + Pemetrexed/Cisplatin (Phase 1) | Axitinib (Continuous) + Pemetrexed/Cisplatin (Phase 2) | Axitinib (Modified) + Pemetrexed/Cisplatin (Phase 2) | Pemetrexed/Cisplatin (Phase 2)
Started | 10 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 10 | 0 | 0 | 0
Not completed — Death | 6 | 0 | 0 | 0
Not completed — Other | 4 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Axitinib + Pemetrexed/Cisplatin (Phase 1) | Axitinib (Continuous) + Pemetrexed/Cisplatin (Phase 2) | Axitinib (Modified) + Pemetrexed/Cisplatin (Phase 2) | Pemetrexed/Cisplatin (Phase 2)
Started | 0 | 55 | 58 | 57
Treated | 0 | 55 | 58 | 55
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 55 | 58 | 57
Not completed — Death | 0 | 37 | 48 | 31
Not completed — Protocol Violation | 0 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1
Not completed — Other | 0 | 1 | 2 | 4
Not completed — Study Terminated by Sponsor | 0 | 13 | 7 | 14
Not completed — Randomized but not treated | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Axitinib + Pemetrexed/Cisplatin (Phase 1) | Axitinib (Continuous) + Pemetrexed/Cisplatin (Phase 2) | Axitinib (Modified) + Pemetrexed/Cisplatin (Phase 2) | Pemetrexed/Cisplatin (Phase 2) | Total
Number analyzed (Participants) | 10 | 55 | 58 | 57 | 180
Age, Customized [Number; unit: participants]
  Less Than 65 Years | 5 | 35 | 34 | 43 | 117
  Greater Than or Equal to 65 Years | 5 | 20 | 24 | 14 | 63
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 21 | 21 | 20 | 63
  Male | 9 | 34 | 37 | 37 | 117

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Time in months from the date of randomization to first documentation of objective tumor progression or death due to any cause. PFS was calculated as (first event date minus minus the date of randomization plus 1) divided by 30.4. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]); death was determined from AE data (where the outcome was "Death") or from the end of study data.
Time Frame: Phase 2 baseline until the date of first documented progression or death due to any cause or initiation of subsequent anticancer therapy, assessed every 6 weeks up to 84 weeks
Population: Full analysis (FA) population, included all participants randomized with study medication assignment designated according to initial randomization, regardless of whether participants received study medication or received a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib (Continuous) + Pemetrexed/Cisplatin (Phase 2) | Axitinib (Modified) + Pemetrexed/Cisplatin (Phase 2) | Pemetrexed/Cisplatin (Phase 2)
Number analyzed (Participants) | 55 | 58 | 57
months | 8.0 [6.7 to 10.0] | 8.1 [6.8 to 9.9] | 7.1 [5.8 to 9.4]
Statistical Analysis 1: Comparison: Axitinib (Continuous) + Pemetrexed/Cisplatin (Phase 2) vs Pemetrexed/Cisplatin (Phase 2); P-value was calculated using 1-sided log rank test, stratified by Eastern Cooperative Oncology Group (ECOG) performance status (0 or 1) and gender (male or female). Hazard ratio (HR): the stratified Cox model was fitted, using the same stratification variables as above; Test type: Superiority or Other; p = 0.3037, Log Rank; One-sided log-rank test at alpha = 0.20 significance level was used; Hazard Ratio (HR) = 0.831, 95% CI 2-sided [0.508 to 1.360]
Statistical Analysis 2: Comparison: Axitinib (Modified) + Pemetrexed/Cisplatin (Phase 2) vs Pemetrexed/Cisplatin (Phase 2); P-value was calculated using 1-sided log rank test, stratified by ECOG performance status (0 or 1) and gender (male or female). HR: the stratified Cox model was fitted, using the same stratification variables as above; Test type: Superiority or Other; p = 0.3565, Log Rank; One-sided log-rank test at alpha = 0.20 significance level was used; Hazard Ratio (HR) = 0.947, 95% CI 2-sided [0.580 to 1.546]

2. Secondary Outcome: Overall Survival (OS)
Description: Time in months from the date of randomization to date of death due to any cause. OS was calculated as (the death date minus the date of randomization plus 1) divided by 30.4. Death was determined from AE data (where outcome was death) or from follow-up contact data (where the participant current status was death).
Time Frame: Baseline until death or collected bimonthly following discontinuation of study treatment until at least 1 year after randomization of the last participant
Population: FA population, included all participants randomized with study medication assignment designated according to initial randomization, regardless of whether participants received study medication or received a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib (Continuous) + Pemetrexed/Cisplatin (Phase 2) | Axitinib (Modified) + Pemetrexed/Cisplatin (Phase 2) | Pemetrexed/Cisplatin (Phase 2)
Number analyzed (Participants) | 55 | 58 | 57
months | 17.0 [12.6 to 22.5] | 14.7 [11.5 to 18.1] | 15.9 [11.1 to NA] — Upper limit of confidence interval (C.I.) was not estimable due to insufficient events as there were few data points.
Statistical Analysis 1: Comparison: Axitinib (Continuous) + Pemetrexed/Cisplatin (Phase 2) vs Pemetrexed/Cisplatin (Phase 2); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.5785, Log Rank; One-sided log-rank test at alpha = 0.20 significance level was used; Hazard Ratio (HR) = 1.046, 95% CI 2-sided [0.648 to 1.690]
Statistical Analysis 2: Comparison: Axitinib (Modified) + Pemetrexed/Cisplatin (Phase 2) vs Pemetrexed/Cisplatin (Phase 2); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.9392, Log Rank; One-sided log-rank test at alpha = 0.20 significance level was used; Hazard Ratio (HR) = 1.449, 95% CI 2-sided [0.919 to 2.285]

3. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with OR based assessment of confirmed complete response (CR)/confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors(RECIST).Confirmed responses: those persist on repeat imaging study at least 4 weeks after initial documentation of response.CR: disappearance of all lesions (target/non target) and no appearance of new lesions.PR: those with at least 30 % decrease in sum of longest dimensions of target lesions taking as reference baseline sum longest dimensions,without progression of non target lesions and no appearance of new lesions.
Time Frame: Phase 2 baseline until the date of first documented progression or discontinuation from the study due to any cause or initiation of subsequent anticancer therapy, assessed every 6 weeks up to 84 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axitinib (Continuous) + Pemetrexed/Cisplatin (Phase 2) | Axitinib (Modified) + Pemetrexed/Cisplatin (Phase 2) | Pemetrexed/Cisplatin (Phase 2)
Number analyzed (Participants) | 55 | 58 | 57
percentage of participants | 45.5 [32.0 to 59.4] | 39.7 [27.0 to 53.4] | 26.3 [15.5 to 39.7]
Statistical Analysis 1: Comparison: Axitinib (Continuous) + Pemetrexed/Cisplatin (Phase 2) vs Pemetrexed/Cisplatin (Phase 2); P-value was calculated using Cochran-Mantel-Haenszel (CMH) test stratified by ECOG performance status (0 or 1) and gender (male or female); Test type: Superiority or Other; p = 0.0143, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.753, 95% CI 2-sided [1.047 to 2.935]
Statistical Analysis 2: Comparison: Axitinib (Modified) + Pemetrexed/Cisplatin (Phase 2) vs Pemetrexed/Cisplatin (Phase 2); P-value was calculated using CMH test stratified by ECOG performance status (0 or 1) and gender (male or female); Test type: Superiority or Other; p = 0.0665, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.512, 95% CI 2-sided [0.870 to 2.626]

4. Secondary Outcome: Duration of Response (DR)
Description: Time in months from the first documentation of objective tumor response to objective tumor progression or death due to any cause, whichever occurs first. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to cause minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 30.4. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: as for outcome 3
Population: Subgroup of participants from the FA population with a confirmed objective tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib (Continuous) + Pemetrexed/Cisplatin (Phase 2) | Axitinib (Modified) + Pemetrexed/Cisplatin (Phase 2) | Pemetrexed/Cisplatin (Phase 2)
Number analyzed (Participants) | 25 | 23 | 15
months | 7.82 [5.6 to 11.4] | 6.73 [5.0 to 7.8] | 7.10 [4.2 to 24.7]

5. Secondary Outcome: Change From Baseline in Monroe Dunaway (MD) Anderson Symptom Inventory (MDASI) Symptom Severity Score
Description: Symptom severity score is comprised of average of 13 MDASI core items (pain, fatigue, nausea, disturbed sleep, distressed, shortness of breath, remembering things, lack of appetite, drowsy, dry mouth, sadness, vomiting, numbness or tingling) and ranges from 0 to 10. Participants were asked to rate severity of each symptom at their worst in last 24 hours; each item rated from 0 to 10, with 0 = symptom not present and 10 = as bad as you can imagine. Lower scores indicated better outcome.
Time Frame: Phase 2 baseline (Cycle1/Day1), Cycle1/Day8, then Day 1 and 8 of each cycle of chemotherapy (C) up to CycleC6, Day 1 of each cycle of single-agent phase (A) up to CycleA8 and end of treatment (EOT)
Population: FA population; 'N' (number of participants analyzed) signifies participants evaluable for this measure and 'n' is number of participants analyzed at specific time point for each treatment arm respectively.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Axitinib (Continuous) + Pemetrexed/Cisplatin (Phase 2) | Axitinib (Modified) + Pemetrexed/Cisplatin (Phase 2) | Pemetrexed/Cisplatin (Phase 2)
Number analyzed (Participants) | 55 | 55 | 53
units on a scale
  Phase 2 baseline (CycleC1/Day 1), (n= 55, 55, 53) | 1.75 [1.32 to 2.18] | 2.09 [1.67 to 2.50] | 1.80 [1.33 to 2.27]
  Change at CycleC1/Day 8, (n= 49, 49, 50) | 1.55 [1.09 to 2.02] | 0.36 [0.00 to 0.72] | 0.95 [0.56 to 1.34]
  Change at CycleC2/Day1 (n= 51, 51, 41) | 0.12 [-0.26 to 0.49] | -0.05 [-0.46 to 0.35] | 0.39 [0.01 to 0.77]
  Change at CycleC2/Day8 (n= 39, 38, 34) | 1.52 [0.98 to 2.06] | 0.39 [-0.14 to 0.92] | 0.69 [0.24 to 1.13]
  Change at CycleC3/Day1 (n= 45, 47, 39) | 0.57 [0.16 to 0.97] | 0.29 [-0.13 to 0.71] | 0.32 [-0.15 to 0.79]
  Change at CycleC3/Day8 (n= 38, 35, 32) | 1.33 [0.75 to 1.92] | 0.87 [0.18 to 1.56] | 1.15 [0.61 to 1.68]
  Change at CycleC4/Day1 (n= 43, 43, 38) | 0.85 [0.28 to 1.42] | 0.48 [-0.06 to 1.02] | 0.37 [-0.05 to 0.79]
  Change at CycleC4/Day8 (n= 33, 33, 27) | 1.37 [0.64 to 2.09] | 0.90 [0.30 to 1.51] | 1.48 [0.77 to 2.19]
  Change at CycleC5/Day1 (n= 35, 34, 29) | 0.59 [0.05 to 1.12] | 0.48 [-0.17 to 1.12] | 0.72 [0.25 to 1.18]
  Change at CycleC5/Day8 (n= 29, 26, 25) | 1.19 [0.38 to 2.00] | 0.82 [0.10 to 1.55] | 1.16 [0.46 to 1.87]
  Change at CycleC6/Day1 (n= 27, 28, 28) | 0.67 [0.04 to 1.30] | 0.42 [-0.22 to 1.06] | 0.67 [0.11 to 1.23]
  Change at CycleC6/Day8 (n= 25, 25, 21) | 1.44 [0.71 to 2.17] | 0.85 [0.23 to 1.47] | 1.28 [0.48 to 2.08]
  Change at CycleA1/Day1 (n= 35, 33, 21) | 0.63 [0.27 to 0.99] | 0.24 [-0.32 to 0.79] | 0.68 [-0.09 to 1.45]
  Change at CycleA2/Day1 (n= 32, 30, 14) | 0.36 [-0.11 to 0.83] | -0.01 [-0.55 to 0.54] | 0.14 [-0.49 to 0.77]
  Change at CycleA3/Day1 (n= 27, 26, 10) | 0.25 [-0.30 to 0.79] | 0.01 [-0.63 to 0.65] | 0.12 [-0.38 to 0.63]
  Change at CycleA4/Day1 (n= 22, 25, 0) | 0.03 [-0.65 to 0.70] | 0.07 [-0.56 to 0.70] | NA [NA to NA] — Data was not summarized because there was insufficient number of participants to calculate change from baseline at visit.
  Change at CycleA5/Day1 (n= 17, 23, 12) | 0.19 [-0.78 to 1.16] | -0.12 [-0.73 to 0.48] | 0.30 [-0.37 to 0.96]
  Change at CycleA6/Day1 (n= 17, 16, 10) | 0.10 [-0.56 to 0.77] | -0.23 [-1.21 to 0.76] | 0.14 [-0.83 to 1.11]
  Change at CycleA7/Day1 (n= 15, 15, 0) | -0.26 [-0.99 to 0.47] | -0.33 [-1.37 to 0.70] | NA [NA to NA] — Data was not summarized because there was insufficient number of participants to calculate change from baseline at visit.
  Change at CycleA8/Day1 (n= 15, 14, 10) | -0.28 [-0.91 to 0.35] | 0.30 [-0.76 to 1.36] | 0.02 [-1.15 to 1.20]
  Change at CycleA9/Day1 (n= 13, 11, 0) | -0.46 [-1.29 to 0.38] | 0.34 [-0.51 to 1.19] | NA [NA to NA] — Data was not summarized because there was insufficient number of participants to calculate change from baseline at visit.
  Change at CycleA10/Day1 (n= 0, 10, 0) | NA [NA to NA] — Data was not summarized because there was insufficient number of participants to calculate change from baseline at visit. | 0.61 [-0.38 to 1.59] | NA [NA to NA] — Data was not summarized because there was insufficient number of participants to calculate change from baseline at visit.
  Change at EOT (n= 40, 35, 31) | 0.66 [0.12 to 1.20] | 1.02 [0.40 to 1.63] | 0.99 [0.33 to 1.64]

6. Secondary Outcome: Change From Baseline in Monroe Dunaway (MD) Anderson Symptom Inventory (MDASI) Symptom Interference Score
Description: Symptom interference score is comprised of average of 6 function items from MDASI core (general activity, mood, work, relations with others, walking, and enjoyment of life) and ranges from 0 to 10. Participants were asked to rate how much symptoms have interfered in last 24 hours; each item rated from 0 to 10, with 0 = did not interfere and 10 = interfered completely. Lower scores indicated better outcome.
Time Frame: Phase 2 baseline (Cycle1/Day1), Cycle1/Day8, then Day 1 and 8 of each cycle of chemotherapy (C) up to CycleC6, Day 1 of each cycle of single-agent phase (A) up to CycleA8 and EOT
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Axitinib (Continuous) + Pemetrexed/Cisplatin (Phase 2) | Axitinib (Modified) + Pemetrexed/Cisplatin (Phase 2) | Pemetrexed/Cisplatin (Phase 2)
Number analyzed (Participants) | 55 | 55 | 53
units on a scale
  Phase 2 baseline (CycleC1/Day 1), (n= 55, 55, 53) | 2.36 [1.64 to 3.08] | 2.97 [2.27 to 3.68] | 2.64 [1.92 to 3.37]
  Change at CycleC1/Day 8, (n= 49, 49, 50) | 1.48 [0.80 to 2.16] | -0.03 [-0.75 to 0.68] | 0.81 [0.27 to 1.36]
  Change at CycleC2/Day1 (n= 51, 51, 41) | 0.27 [-0.21 to 0.75] | -0.24 [-0.76 to 0.29] | 0.30 [-0.25 to 0.84]
  Change at CycleC2/Day8 (n= 39, 38, 34) | 2.00 [1.07 to 2.93] | 0.03 [-0.61 to 0.66] | 0.52 [0.05 to 0.99]
  Change at CycleC3/Day1 (n= 45, 47, 39) | 0.64 [0.07 to 1.21] | -0.21 [-0.81 to 0.40] | 0.03 [-0.41 to 0.46]
  Change at CycleC3/Day8 (n= 38, 35, 32) | 1.54 [0.57 to 2.50] | 0.28 [-0.46 to 1.03] | 0.41 [-0.00 to 0.82]
  Change at CycleC4/Day1 (n= 43, 43, 38) | 0.72 [-0.18 to 1.62] | 0.11 [-0.50 to 0.73] | 0.28 [-0.16 to 0.71]
  Change at CycleC4/Day8 (n= 33, 33, 27) | 1.39 [0.20 to 2.58] | 1.08 [0.23 to 1.92] | 1.20 [0.48 to 1.93]
  Change at CycleC5/Day1 (n= 35, 34, 29) | 0.14 [-0.67 to 0.95] | -0.05 [-0.88 to 0.78] | 0.49 [-0.10 to 1.09]
  Change at CycleC5/Day8 (n= 29, 26, 25) | 0.78 [-0.42 to 1.97] | 0.88 [-0.19 to 1.94] | 0.76 [-0.03 to 1.55]
  Change at CycleC6/Day1 (n= 27, 28, 28) | 0.18 [-0.76 to 1.12] | 0.17 [-0.68 to 1.01] | 0.66 [-0.04 to 1.36]
  Change at CycleC6/Day8 (n= 25, 25, 21) | 1.00 [-0.16 to 2.16] | 1.04 [0.17 to 1.91] | 1.20 [0.32 to 2.08]
  Change at CycleA1/Day1 (n= 35, 33, 21) | 0.49 [-0.20 to 1.18] | 0.39 [-0.34 to 1.13] | 0.96 [0.28 to 1.64]
  Change at CycleA2/Day1 (n= 32, 30, 14) | 0.25 [-0.52 to 1.02] | 0.16 [-0.67 to 0.98] | 0.10 [-0.82 to 1.01]
  Change at CycleA3/Day1 (n= 27, 26, 10) | 0.02 [-0.82 to 0.87] | -0.20 [-1.15 to 0.76] | 0.27 [-0.43 to 0.96]
  Change at CycleA4/Day1 (n= 22, 25, 0) | 0.33 [-0.43 to 1.10] | 0.23 [-0.58 to 1.05] | NA [NA to NA] — Data was not summarized because there was insufficient number of participants to calculate change from baseline at visit.
  Change at CycleA5/Day1 (n= 17, 23, 12) | 0.36 [-0.54 to 1.27] | 0.12 [-1.02 to 1.27] | 0.40 [-0.56 to 1.37]
  Change at CycleA6/Day1 (n= 17, 16, 10) | 0.16 [-0.47 to 0.79] | 0.28 [-0.82 to 1.39] | 0.12 [-0.92 to 1.15]
  Change at CycleA7/Day1 (n= 15, 15, 0) | 0.12 [-0.68 to 0.92] | 0.00 [-1.14 to 1.15] | NA [NA to NA] — Data was not summarized because there was insufficient number of participants to calculate change from baseline at visit.
  Change at CycleA8/Day1 (n= 15, 14, 10) | -0.07 [-0.96 to 0.82] | 0.30 [-0.70 to 1.29] | 0.42 [-0.39 to 1.23]
  Change at CycleA9/Day1 (n= 13, 11, 0) | -0.13 [-1.03 to 0.77] | 1.05 [0.09 to 2.00] | NA [NA to NA] — Data was not summarized because there was insufficient number of participants to calculate change from baseline at visit.
  Change at CycleA10/Day1 (n= 0, 10, 0) | NA [NA to NA] — Data was not summarized because there was insufficient number of participants to calculate change from baseline at visit. | 1.03 [0.06 to 2.01] | NA [NA to NA] — Data was not summarized because there was insufficient number of participants to calculate change from baseline at visit.
  Change at EOT (n= 40, 35, 31) | 0.69 [-0.26 to 1.64] | 0.69 [-0.22 to 1.59] | 0.91 [0.06 to 1.77]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Axitinib + Pemetrexed/Cisplatin (Phase 1) | Axitinib (Continuous) + Pemetrexed/Cisplatin (Phase 2) | Axitinib (Modified) + Pemetrexed/Cisplatin (Phase 2) | Pemetrexed/Cisplatin (Phase 2)
Serious Adverse Events (participants affected / at risk) | 1/10 | 19/55 | 20/58 | 13/55
Other Adverse Events (participants affected / at risk) | 10/10 | 54/55 | 56/58 | 54/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib + Pemetrexed/Cisplatin (Phase 1) (N=10) | Axitinib (Continuous) + Pemetrexed/Cisplatin (Phase 2) (N=55) | Axitinib (Modified) + Pemetrexed/Cisplatin (Phase 2) (N=58) | Pemetrexed/Cisplatin (Phase 2) (N=55)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 4 | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestine ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 5 | 2 | 2
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 2
Fatigue (General disorders) | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 1 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 3 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 2 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 1
Post thrombotic syndrome (Vascular disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Femoral artery occlusion (Vascular disorders) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Basal ganglia infarction (Nervous system disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib + Pemetrexed/Cisplatin (Phase 1) (N=10) | Axitinib (Continuous) + Pemetrexed/Cisplatin (Phase 2) (N=55) | Axitinib (Modified) + Pemetrexed/Cisplatin (Phase 2) (N=58) | Pemetrexed/Cisplatin (Phase 2) (N=55)
Anaemia (Blood and lymphatic system disorders) | 5 | 7 | 19 | 23
Leukopenia (Blood and lymphatic system disorders) | 1 | 6 | 8 | 3
Neutropenia (Blood and lymphatic system disorders) | 5 | 17 | 12 | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 8 | 4 | 3
Hypoacusis (Ear and labyrinth disorders) | 0 | 3 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 3 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 9 | 4 | 5
Abdominal pain upper (Gastrointestinal disorders) | 1 | 5 | 8 | 7
Cheilitis (Gastrointestinal disorders) | 0 | 4 | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 20 | 15 | 23
Diarrhoea (Gastrointestinal disorders) | 5 | 22 | 20 | 9
Flatulence (Gastrointestinal disorders) | 0 | 4 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 3 | 2 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 4 | 3 | 3
Nausea (Gastrointestinal disorders) | 6 | 37 | 30 | 32
Stomatitis (Gastrointestinal disorders) | 0 | 10 | 7 | 3
Vomiting (Gastrointestinal disorders) | 4 | 26 | 19 | 14
Asthenia (General disorders) | 5 | 9 | 11 | 7
Chest pain (General disorders) | 1 | 6 | 6 | 5
Fatigue (General disorders) | 8 | 27 | 25 | 25
Oedema (General disorders) | 0 | 4 | 2 | 4
Oedema peripheral (General disorders) | 0 | 3 | 6 | 3
Pain (General disorders) | 0 | 3 | 6 | 2
Pyrexia (General disorders) | 0 | 5 | 10 | 3
Nasopharyngitis (Infections and infestations) | 0 | 9 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 3 | 3 | 1
Blood creatinine increased (Investigations) | 2 | 5 | 2 | 3
Blood thyroid stimulating hormone increased (Investigations) | 0 | 4 | 2 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 4 | 3 | 3
Neutrophil count decreased (Investigations) | 0 | 5 | 2 | 1
Weight decreased (Investigations) | 1 | 4 | 6 | 4
Decreased appetite (Metabolism and nutrition disorders) | 7 | 29 | 28 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 7 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4 | 4 | 0
Dizziness (Nervous system disorders) | 0 | 4 | 6 | 3
Dysgeusia (Nervous system disorders) | 2 | 9 | 6 | 1
Headache (Nervous system disorders) | 2 | 12 | 17 | 9
Neuropathy peripheral (Nervous system disorders) | 1 | 5 | 2 | 1
Depression (Psychiatric disorders) | 2 | 4 | 4 | 0
Insomnia (Psychiatric disorders) | 0 | 13 | 8 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 12 | 7 | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 13 | 8 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 13 | 13 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 8 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 8 | 5 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 4 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 9 | 6 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 5 | 3 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 10 | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 4 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 7 | 10 | 5
Hypertension (Vascular disorders) | 7 | 37 | 28 | 6
Hypotension (Vascular disorders) | 0 | 6 | 4 | 3
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 2 | 3 | 2
Lacrimation increased (Eye disorders) | 2 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 2 | 0 | 3
Dry eye (Eye disorders) | 0 | 0 | 3 | 0
Vision blurred (Eye disorders) | 0 | 2 | 2 | 3
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 3 | 2
Aerophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 2 | 4 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 3 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 5 | 4
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophageal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Perianal erythema (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal tenesmus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 3 | 0
Face oedema (General disorders) | 0 | 1 | 1 | 3
Mucosal inflammation (General disorders) | 1 | 2 | 4 | 3
Cyst (General disorders) | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Mucous membrane disorder (General disorders) | 1 | 0 | 0 | 0
Xerosis (General disorders) | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 3 | 3
Sinusitis (Infections and infestations) | 0 | 1 | 3 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 1
Aspartate aminotransferase (Investigations) | 1 | 0 | 0 | 0
Blood creatinine (Investigations) | 1 | 0 | 0 | 0
Haemoglobin (Investigations) | 1 | 0 | 0 | 0
Hypophonesis (Investigations) | 1 | 0 | 0 | 0
Neutrophil count (Investigations) | 1 | 0 | 0 | 0
Transaminases (Investigations) | 1 | 0 | 0 | 0
White blood cell count (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 3 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 2 | 2 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1 | 4 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 7 | 3 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 1 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 0 | 3 | 0
Paraesthesia (Nervous system disorders) | 2 | 2 | 5 | 3
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 5 | 0
Agitation (Psychiatric disorders) | 2 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 3
Expressive language disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 3 | 1 | 7 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal pain (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 2 | 3 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 3 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 2 | 4
Alanine aminotransferase increased (Investigations) | 0 | 0 | 3 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.